CLINICAL TRIAL: NCT05191264
Title: Combination of Percutaneous Screw Fixation and Cementoplasty for Lytic Bone Metastases: Feasibility, Safety and Early Clinical Outcomes. Monocentric Study
Brief Title: Combination of Percutaneous Screw Fixation and Cementoplasty for Lytic Bone Metastases
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN942019/CHUSTE
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Interventional Radiology
Keywords: Screw fixation; cementoplasty; interventional radiology; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- percutaneous osteosynthesis and cementoplasty procedure: Patient with percutaneous osteosynthesis and cementoplasty procedure will be included.
  Patients have assessed for pain and quality of life during consultations as part of an interventional radiology procedure (pre-procedure consultation, and follow-up consultations at 1, 3, 6 and 12 months after the procedure.
  Interventions: Other: EQ5D (EuroQol 5 Dimensions); Other: Numerical Rating Scale (NRS); Other: evaluated the consumption of analgesics

INTERVENTIONS:
Other: EQ5D (EuroQol 5 Dimensions) — The evaluation of the quality of life was conducted with the EQ5D (EuroQol 5 Dimensions) score (min 0: bad health and max:100 good health).
  Other Names: evaluation of the quality of life
Other: Numerical Rating Scale (NRS) — the type and intensity of pain will be evaluated by Numerical Rating Scale (NRS) from 0 to 10 in different positions and in different activities (e.g. background pain, general maximum/minimum pain, pain of the site treated by the procedure, pain at rest, in lying position, in sitting position, in standing position, at bearing weight, in walking, description of painful irradiations, nocturnal awakenings).
  Other Names: evaluation of the type and intensity of pain
Other: evaluated the consumption of analgesics — the consumption of analgesics by step and by dosage will be evaluated.

SUMMARY:
In oncology, therapeutic progress has allowed a significant increase in life-expectancy: a growing number of cancer survivors live to more advanced metastatic stages. Consequently, the prevalence of secondary bone lesions is increasing, which are frequent and disabling. They are responsible for pain and a high risk of pathological fractures. The average prevalence of pain in cancer represents 53% for all stages combined and 64% for metastatic stages.

Analgesics, radiotherapy and surgery are widely used in this context, but are not without side effects.

Cementoplasty is an interventional radiology procedure that has improved the palliative management of bone lesions. It consists of a percutaneous injection of polymethylmethacrylate-based cement, whose physical and chemical properties provide resistance to compressive stress during weight-bearing activities. However, one of the main disadvantages of cement is its low resistance to torsional stress, as evidenced notably in vitro tests. Thus, cementoplasty alone is very effective at the spinal level (compressive forces) to reduce pain and risk of fracture, but much less effective at the level of other bones that are subjected to torsional stresses, notably the pelvis and femur (40% fracture rate at one year after cementoplasty alone of femoral metastasis).

Fixation using a combination of metal screws and cement provides resistance to torsional and compressive stress. In addition, it has been shown that there is a significant risk of secondary screw displacement if screws are not combined with cement in secondary bone lesions. Combination of percutaneous screw fixation and cementoplasty is a mini-invasive procedure which allows limiting complications and the duration of treatment: early standing up, almost no blood loss, reduced risk of venous thromboembolism (VTE), rapid healing.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate feasibility, safety, and efficacy of combination of percutaneous screw fixation and cementoplasty for lytic bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* patients who received osteosynthesis/cementoplasty for Lytic Bone Metastases

Exclusion Criteria:

* patient's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with percutaneous osteosynthesis and cementoplasty procedure will be included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of the procedure (Yes or No) | Just after the end of the procedure
  The technical success of the procedure is defined as (all criteria have to be fulfilled) :
  * the correct placement of the screw(s),
  * any complication as major cement leakage such as intra-articular or intra-vascular leakage, abundant bleeding, vascular or nervous lesion, displacement of bone fragment
  Theses criteria are measured on CT-scan

SECONDARY OUTCOMES:
Adverse events | Months: 1, 3, 6 and 12
  To confirm the safety of the procedure, all adverse events related to the procedure are screened and reported
Numerical Rating Scale | Months: 1, 3, 6 and 12
  Numerical Rating Scale (NRS) evaluates the pain. This scale starts from 0 (no pain) to 10 (maximal pain)
EuroQol 5 Dimensions (EQ5D) | Months: 1, 3, 6 and 12
  EQ5D evaluates the quality of life.. Patients are asked to describe their own health and also provide a self-rating on a 20-cm vertical scale with endpoints of 'best imaginable health state' set at 100 and 'worst imaginable health state' set at 0
Consumption of opioids (mg/day) | Months: 1, 3, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No